CLINICAL TRIAL: NCT07112300
Title: Evaluation of the Efficacy of Ultrasound-guided Cervical Root Pulsed Radiofrequency Treatment at the Intertubercular and Interscalene Levels in the Treatment of Cervical Radicular Pain
Brief Title: Interscalene and ıntertuberculary Pulsed Radiofrequency for Cervical Radiculopathy
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, medical doctor, Diskapi Teaching and Research Hospital
Other Study IDs: Interscalene pRF
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cervical Radicular Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interscalene cervical nerve radiofrequency: The group treated with interscalene pulsed radiofrequency intervention
  Interventions: Procedure: cervical nerve radiofrequency
- Intertubercular cervical nerve radiofrequency: The group was treated with intertubercular pulsed radiofrequency intervention
  Interventions: Procedure: cervical nerve radiofrequency

INTERVENTIONS:
Procedure: cervical nerve radiofrequency — Pulsed radiofrequency treatment is applied to the cervical 5-6-7 nerve roots defined under ultrasound guidance in the intertubercular or interscalene space by approaching the cervical 5-6-7 nerve roots with an inplane technique via a cannula electrode.

SUMMARY:
This study examines the different application techniques of ultrasound-guided pulsed radiofrequency treatment of cervical spinal nerves for cervical radicular pain.

Patients with radiologic imaging findings of C5-C6-C7 disc protrusion or extrusion, with compatible clinical and physical examinations and who have undergone ultrasound-guided spinal cervical nerve radiofrequency treatment in our clinic will be evaluated. Patients' background information will be taken in their files and missing information will be completed by phone call. Pain scores at 3 and 6 months after the procedure will be recorded by scoring from 1 to 10. Patients will not undergo any interventional procedure for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically proven extruded/protruded discopathy at C5/C6/C7 levels
* Presence of radicular pain that can be provoked by physical examination
* Consistent with radiologic imaging findings.

Exclusion Criteria:

* No surgical procedures in the cervical region
* Concomitant pregnancy, malignancy, bleeding diathesis
* Presence of rheumatologic diseases associated with concomitant chronic pain syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical radicular neuropathic pain
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Visual Analouge Scale | pretreatment, 3.- 6. months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.

SECONDARY OUTCOMES:
Neck Disability Index | pretreatment, 6. months
  Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided